CLINICAL TRIAL: NCT01590147
Title: Supportive Intervention Programs to Lessen Treatment Related Symptoms
Brief Title: Supportive Intervention Programs Study
Acronym: SIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00016716; NCI-2011-01093 (Registry Identifier: NCI); CCCWFU 98211 (Other: NCI)
Record Dates: First submitted 2012-05-01; First posted 2012-05-02 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Fatigue; Nausea and Vomiting; Pain; Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage I-IVB Colon Cancer; Stage I-IVB Rectal Cancer
MeSH Terms: conditions — Fatigue; Nausea; Vomiting; Pain; Colonic Neoplasms; Rectal Neoplasms | interventions — Yoga; Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (YST) (Experimental): Patients participate in three 15-minute YST sessions, comprising awareness meditation practice, movement practice, and breathing practice and relaxation. Patients also receive a CD recording of a 15-minute YST session and are instructed to practice the YST at home 4 times weekly.
  Interventions: Procedure: Yoga therapy; Other: questionnaire administration; Procedure: quality-of-life assessment; Other: laboratory biomarker analysis; Other: assessment of therapy complications; Procedure: management of therapy complications
- Arm 2 (CE) (Active Comparator): Patients participate in three 15-minute CE sessions, comprising empathic attention with an interventionist who allows patients to direct the flow of conversation and provides supportive comments according to standardized procedures. Patients also receive CDs with recorded information related to coping with colorectal cancer similar in length to the suggested practice time in Arm I.
  Interventions: Other: questionnaire administration; Procedure: quality-of-life assessment; Other: laboratory biomarker analysis; Other: assessment of therapy complications; Procedure: management of therapy complications; Other: educational intervention

INTERVENTIONS:
Procedure: Yoga therapy — receive YST
  Arms: Arm 1 (YST)
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
Other: laboratory biomarker analysis — Correlative studies
Other: assessment of therapy complications — Ancillary studies
Procedure: management of therapy complications — Receive YST or CE
  Other Names: complications of therapy, management of
Other: educational intervention — Receive CE
  Arms: Arm 2 (CE)

SUMMARY:
This randomized clinical trial studies the preliminary efficacy of a yoga skills training (YST) compared to counseling and education (CE) for reducing treatment-related symptoms in patients with colorectal cancer who are receiving chemotherapy. The YST may reduce fatigue, other treatment-related symptoms, and improve the quality of life (QOL) of patients with colorectal cancer. It is not yet known whether YST is more effective then CE in reducing these outcomes.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To establish the feasibility of implementing a YST among patients undergoing chemotherapy. This includes the feasibility of implementing yoga in a treatment setting, and patient recruitment, adherence, and retention.

II. To obtain preliminary data on the efficacy of a YST for reducing fatigue among patients undergoing chemotherapy.

III. To obtain exploratory data on the impact of a YST on other treatment-related symptoms (e.g., pain, distress, nausea) and QOL.

IV. To obtain exploratory data on the impact of a YST on potential psychological (self-efficacy for coping with cancer, response expectancies for symptoms) and physiological (interleukin [IL]-6 [IL-6], IL-1 Receptor Antagonist [IL-1Ra], tumor necrosis factor- alpha [TNF-a], soluble TNF receptor I [sTNFRI], C-reactive protein [CRP]) mediators that may explain the impact of the YST on fatigue.

OUTLINE: Patients (n=20) are randomized to 1 of 2 treatment arms.

ARM I: Patients participate in three 15-minute YST sessions, comprising awareness meditation practice, movement practice, and breathing practice and relaxation. Patients also receive a compact disc (CD) recording of a 15-minute YST session and are instructed to practice the YST at home 4 times weekly.

ARM II: Patients participate in three 15-minute CE sessions, comprising empathic attention with an interventionist who allows patients to direct the flow of conversation and provides supportive comments according to standardized procedures. Patients also receive CDs with recorded information related to coping with colorectal cancer similar in length to the suggested practice time in Arm I.

The interventions (Week 2, Week 4, Week 6) and assessments (Week 0, Week 4, Week 8) are implemented during visits for chemotherapy (every two weeks).

ELIGIBILITY:
Inclusion Criteria:

* Signed protocol specific informed consent
* Are diagnosed with colorectal cancer
* Recruited within 2 weeks of initiating chemotherapy (including reinitiating chemotherapy after a treatment holiday of greater than or equal to 4 weeks)
* Able to understand written and spoken English

Exclusion Criteria:

* Under age 18 (children with colorectal cancer)
* Unable to read or understand English
* Vulnerable subjects (except those who are economically or educationally disadvantaged)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing a YST among patients undergoing chemotherapy (participating rate, adherence, and retention) | Up to 8 weeks
  The proportion of participants who participated in all study sessions and those who completed all assessments will be computed and compared by demographic characteristics and intervention group. The investigators will model the relationship between adherence and baseline scores of the measures, as well as change in scores.

SECONDARY OUTCOMES:
Preliminary efficacy of YST, in terms of reducing fatigue | At week 8
  Measured by the Functional Assessment of Cancer Therapy - Fatigue (FACT-F) subscale. Assessed using analysis of covariance (ANCOVA) models, accounting for possible confounding variables (e.g., medication use) from baseline to post intervention.
Treatment related symptoms and QOL | At week 8
  The Functional Assessment of Cancer Therapy- Colorectal (FACT-C; 37) will be used to evaluate overall QOL (physical, social, emotional, and functional well-being) and colorectal cancer specific symptoms (e.g., cramps in stomach, control of bowels). Assessed using ANCOVA.
Mediating variables (self efficacy, response expectancies, inflammatory biomarkers) intervention effect on fatigue, treatment-related symptoms, and QOL | Up to 8 weeks
  Assessed using a simultaneous model of the mediators and the intervention effect in the ANCOVA model.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie J Sohl, PhD, Principal Investigator — Wake Forest
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States